CLINICAL TRIAL: NCT07162285
Title: Efficacy of Delivery Room Bubble Continuous Positive Airway Pressure in Preterm Neonates <34 Weeks Having Respiratory Distress
Brief Title: "Effectiveness of Delivery Room Bubble CPAP in Preterm Infants With Respiratory Distress
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Nuzhat Nuary Jui, Resident Doctor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4724
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: Delivery Room Bubble CPAP
  Supplemental Oxygen (control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delivery Room Bubble CPAP (Experimental): Preterm neonates (<34 weeks gestation) with respiratory distress will receive bubble continuous positive airway pressure (bCPAP) initiated in the delivery room within 10 minutes of birth. The intervention will be delivered via nasal prongs with pressure settings titrated as per institutional protocol. The aim is to provide continuous distending pressure to stabilize alveoli, improve oxygenation, and reduce the need for intubation, surfactant, and mechanical ventilation.
  Interventions: Device: Delivery Room Bubble CPAP
- Delivery Room Supplemental Oxygen (Active Comparator): Preterm neonates (<34 weeks gestation) with respiratory distress will receive supplemental oxygen therapy in the delivery room within 10 minutes of birth, administered by standard delivery methods (e.g., mask and oxygen flow). This group will serve as the comparator to evaluate whether early initiation of bubble CPAP improves respiratory outcomes compared to oxygen alone.
  Interventions: Other: Delivery Room Supplemental Oxygen

INTERVENTIONS:
Device: Delivery Room Bubble CPAP — delivery room bubble CPAP initiated within 10 minutes of birth for preterm neonates <34 weeks, using water-seal oscillation system via nasal prongs.
  Arms: Delivery Room Bubble CPAP
Other: Delivery Room Supplemental Oxygen — Standard oxygen therapy initiated within 10 minutes of birth via mask/tubing, without positive pressure support.
  Arms: Delivery Room Supplemental Oxygen

SUMMARY:
Background

When babies are born too early (preterm), their lungs are often not fully developed. They may have trouble breathing because their airways and chest are not strong enough, and their lungs don't make enough surfactant (a natural substance that keeps the lungs open). This makes their tiny lungs collapse easily, causing breathing problems.

Continuous Positive Airway Pressure (CPAP) is a safe and gentle way to help these babies breathe. CPAP works by sending a steady flow of air into the baby's nose, which keeps the lungs open and helps the baby breathe without needing a breathing machine (ventilator). The earlier CPAP is started after birth, the better it may help babies breathe more easily and reduce serious lung problems.

Purpose of the Study

This study will look at whether giving bubble CPAP to preterm babies immediately in the delivery room (within the first 10 minutes after birth) can lower the risk of breathing problems and death during their hospital stay.

How the Study Will Be Done

The research will take place at Bangabandhu Sheikh Mujib Medical University (BSMMU) in Dhaka.

Babies born before 34 weeks of pregnancy who meet the study criteria will be included, with their parents' consent.

Babies will be randomly divided into two groups:

CPAP group - babies will be given bubble CPAP soon after birth in the delivery room.

Control group - babies will receive only oxygen support in the delivery room.

Both groups will then be moved to the Neonatal Intensive Care Unit (NICU) for further treatment as per hospital guidelines.

The results will be compared to see which group had better outcomes.

Expected Outcome

We expect that starting bubble CPAP very early will help preterm babies breathe better, reduce the need for ventilators, and lower the risk of long-term breathing problems or death.

DETAILED DESCRIPTION:
Preterm birth remains one of the most significant contributors to neonatal morbidity and mortality worldwide. Globally, an estimated 15 million infants are born prematurely each year, with the majority occurring in low- and middle-income countries (Blencowe et al., 2013; WHO, 2018). Complications related to prematurity account for over one million deaths annually, and in Bangladesh, prematurity is responsible for nearly one-third of neonatal deaths. Effective respiratory support strategies are therefore critical in improving outcomes in this population.

Continuous Positive Airway Pressure (CPAP) is a well-established mode of non-invasive respiratory support that has been shown to reduce ventilator dependence and the risk of chronic lung disease in preterm infants with respiratory distress. By providing a continuous distending pressure, CPAP stabilizes the alveoli, reduces atelectasis, conserves endogenous surfactant, improves lung compliance, and decreases the work of breathing. These physiological benefits reduce the need for intubation, mechanical ventilation, and exogenous surfactant therapy, all of which are associated with short- and long-term complications.

Bubble CPAP (bCPAP) represents a simple, low-cost, and effective CPAP system particularly suitable for use in resource-limited settings. The system can be assembled using readily available components, and healthcare workers can be trained in its use with relative ease. Compared to ventilator-driven CPAP, bCPAP requires less technical infrastructure and is associated with a lower risk of complications. Previous studies have demonstrated that early initiation of bCPAP is associated with reduced need for intubation and surfactant therapy, shorter duration of respiratory support, and improved weight gain, without increasing adverse outcomes such as pneumothorax (Narendran et al., 2013; Bahareh et al., 2013).

There is increasing evidence that the timing of CPAP initiation plays an important role in determining outcomes. Early initiation of CPAP in the delivery room, before the onset of severe atelectasis, appears more effective than delayed initiation. A systematic review and meta-analysis comparing early versus late CPAP demonstrated that early initiation significantly reduced subsequent use of mechanical ventilation (RR 0.55; 95% CI 0.32-0.96), though effects on mortality, bronchopulmonary dysplasia (BPD), and pneumothorax were not significant (Gupta et al., 2015).

Despite this evidence, there is limited research evaluating the efficacy of immediate delivery room initiation of bCPAP in low-resource countries such as Bangladesh, where the burden of prematurity is high and access to advanced ventilatory support is limited. This randomized controlled trial aims to address this gap.

Study Design and Setting

This is a single-center, randomized controlled clinical trial conducted at Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Bangladesh, involving both the Department of Neonatology and the Department of Obstetrics & Gynecology. The study duration is 18 months, following approval by the Institutional Review Board (IRB).

Eligible preterm neonates (<34 weeks gestation) presenting with respiratory distress at birth will be randomized within 10 minutes of delivery to one of two intervention arms:

Delivery Room bCPAP Group - neonates will receive bubble CPAP initiated in the delivery room.

Control Group - neonates will receive standard oxygen therapy in the delivery room.

Block randomization will be used to ensure equal distribution of participants. Following stabilization, all neonates will be transferred to the Neonatal Intensive Care Unit (NICU) with their assigned respiratory support continued. Subsequent management will follow institutional protocols.

Study Procedures

Upon delivery, eligible neonates will be placed under a radiant warmer. A pulse oximeter will be applied, and respiratory distress will be assessed using a standardized scoring system. In the intervention arm, bCPAP will be initiated using nasal prongs, with pressures titrated according to clinical need. In the control arm, supplemental oxygen will be administered via standard delivery methods.

Daily monitoring will include clinical assessment, oxygen saturation, need for escalation of respiratory support, episodes of apnea, and complications such as pneumothorax, necrotizing enterocolitis, intraventricular hemorrhage, and patent ductus arteriosus. Data will be collected for the first 7 days of life or until discharge, whichever occurs earlier.

Sample Size

Based on prior studies (Desai et al., 2017), an outcome rate of 30% was assumed in the intervention group and 67% in the control group. With α = 0.05 and 80% power, the calculated sample size was 25 participants per group. Allowing for 20% attrition, the final estimated enrollment is 60 neonates.

Statistical Analysis

Data will be analyzed using SPSS version 25. Continuous variables will be summarized as mean ± standard deviation or median (interquartile range) depending on distribution. Categorical variables will be presented as frequencies and percentages. Between-group comparisons will be made using the Student's t-test or Mann-Whitney U test for continuous variables and the chi-square test for categorical variables. Logistic regression will be used to adjust for potential confounders. Statistical significance will be set at p < 0.05. Additional analyses will include correlation testing and ROC curve analysis for predictive variables.

Ethical Considerations

The study will adhere to the principles of the Declaration of Helsinki. Written informed consent will be obtained from parents or guardians prior to enrollment. Data will be de-identified, securely stored, and used exclusively for research purposes. No additional risks are anticipated beyond standard neonatal care.

Significance

This trial is designed to provide robust evidence on the role of early delivery room initiation of bubble CPAP in improving respiratory outcomes for preterm infants in a resource-limited setting. By evaluating both efficacy and safety, the findings are expected to inform national and regional neonatal care strategies, promote scale-up of bCPAP technology, and contribute to reductions in neonatal morbidity and mortality associated with prematurity.

ELIGIBILITY:
Inclusion Criteria:

Neonate gestational age less than 34 weeks delivered at BSMMU. Having respiratory distress.

Exclusion Criteria:

* Congenital anomaly such as cleft lip, cleft palate, congenital diaphragmatic hernia.
* Newborn required delivery room intubation

Ages: 5 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Need for mechanical ventilation | From birth until 7 completed days of life
  This outcome will allow assessment of whether delivery room bubble CPAP reduces respiratory complications with standard supplemental oxygen.
Requirement for surfactant therapy | From birth until 7 completed days of life
  This outcome will allow assessment of whether delivery room bubble CPAP reduces need for surfcatant with standard supplemental oxygen.
Death within the early neonatal period | From birth until 7 completed days of life
  This outcome will allow assessment of whether delivery room bubble CPAP reduces early mortality compared with standard supplemental oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Nuzhat Nuary, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Nuzhat nuary Jui, Dhaka, Bangladesh

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT07162285/Prot_SAP_ICF_000.pdf